CLINICAL TRIAL: NCT05181553
Title: Unravelling the Impact of Diet on Cardiovascular Health in Heterozygous Familial Hypercholesterolemia: a Metabolomic Approach.
Brief Title: Unravelling the Impact of Diet on Cardiovascular Health in Heterozygous Familial Hypercholesterolemia.
Acronym: FH-Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Jean-Philippe Drouin-Chartier, Professor, Laval University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: FH-Diet
Record Dates: First submitted 2021-11-08; First posted 2022-01-06 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Familial Hypercholesterolemia; Nutrition, Healthy; Cholesterol, Elevated; Cholesterol; Metabolic Disorder; Cardiovascular Diseases
Keywords: familial hypercholesterolemia; diet; LDL-cholesterol; metabolome; cardiovascular disease
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Hypercholesterolemia; Metabolic Diseases; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: The proposed research will combine a dietary RCT (objectives 1, 2) and a cohort investigation (objective 3). The dietary intervention will be undertaken as a crossover RCT at the INAF (Université Laval) in Quebec City. Men and women with genetically-defined HeFH will consume in a random order a fully-controlled whole-food plant-based diet low in red and processed meats and high in plant foods (WFPB diet in further sections), and a standard North American diet (SAD diet; i.e. control diet), for 4 weeks each, and separated by a 4-week washout period. The first and second objective consist respectively to investigate the impact of a WFPB diet in place of a SAD on LDL-C concentrations and plasma metabolome.
  The third objective consist to evaluate the association between the plasma metabolomic signature of a diet low in red and processed meats and high in plant foods and cardiovascular disease risk.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Subjects cannot be blinded to treatment allocation, but all laboratory analyses and outcomes will be assessed in a blinded fashion by research staff until the final analyses of the primary outcome are completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Whole-food plant-based diet (WFPB diet) (Experimental): During 28 days, participants will receive the WFPB diet. The WFPB diet emphasizes low intakes of red and processed meats and high intakes of whole plant-based foods with water as the drink of choice, as per Canada's Food Guide. The number of portions of protein foods, whole-grains, fruits and vegetables to be served daily reflects the recommended ¼-¼-½ proportions. Regarding protein quality, vegetable proteins are served more often than animal proteins as stated in Canada's Food Guide. Weekly, red meat is served once and two days are meatless.
  Interventions: Other: Whole-food plant based diet (WFPB diet)
- Standard North American diet (SAD diet) (Experimental): During 28 days, participants will receive the SAD diet. The SAD diet reflects current dietary intakes of the French-Canadian adult population in terms of foods, nutrients, and diet quality, as characterized in recent surveys conducted in an age- and a sex-representative sample of adults from the Province of Quebec. Intakes of whole fruits and vegetables will be low; animal proteins, mostly red and processed meats, will be consumed more often than vegetable proteins; grains will be mostly refined; and ready-to-eat/ready-to-heat foods and sugary beverages will be served daily.
  Interventions: Other: Standard North American diet (SAD diet)

INTERVENTIONS:
Other: Whole-food plant based diet (WFPB diet) — 28-day fully controlled dietary intervention during which participants will receive a whole food plant-based diet that reflects the recommendations of Canada's Food Guide.
  Arms: Whole-food plant-based diet (WFPB diet)
Other: Standard North American diet (SAD diet) — 28-day fully controlled dietary intervention during which participants will receive a diet that reflects the eating habits of Canadians.
  Arms: Standard North American diet (SAD diet)

SUMMARY:
The investigators will first conduct a fully controlled dietary randomized crossover trial (RCT) including 50 adults with HeFH to investigate the impact of a whole food plant-based (WFPB) diet low in red and processed meats and high in plant foods, reflecting Canada's Food Guide, in place of a standard North-American diet on LDL-cholesterol (LDL-C) levels and the plasma metabolome. Such a robust design will also lead to the identification an objective proxy to healthy diet adherence: the metabolomic signature. Secondly, by leveraging a cross-sectional cohort of adults with HeFH, the investigators will evaluate the relationship between the metabolomic signature of the healthy diet and cardiovascular disease risk factors in HeFH.

DETAILED DESCRIPTION:
The research combines a dietary RCT (objectives 1, 2) and a cohort investigation (objective 3), both including adults with genetically-defined HeFH.

The dietary intervention will be undertaken as a crossover RCT at the Institute on nutrition and functional foods (INAF, Laval University) in Quebec City. Participants (men and women with genetically-defined HeFH) will consume in a random order a fully-controlled whole food plant-based diet low in red and processed meats and high in plant foods, reflecting Canada's Food Guide principles (WFPB diet in further sections), and a standard North American diet (SAD diet; i.e. control diet), reflecting current dietary intakes of French-Canadians, for 4 weeks each, and separated by a 4-week washout period.

Once enrolled, participants will enter a 4-week run-in period at the beginning of which they will stop taking their lipid-lowering medication for the study duration (16 weeks). Other medications (e.g. anti-hypertensive drugs, oral contraceptives) will be allowed, but doses will have to remain constant during the study. At the end of the run-in, participants will provide a blood sample and complete a self-administered, validated web-based food-frequency questionnaire. Participants will be randomly assigned to either the WFPB-SAD or SAD-WFPB diet sequence, using a computer-assisted program. The randomization (1:1) will be stratified by sex (female vs male) and LDL-receptor (LDLR) genotype (receptor-negative vs others) in 8 blocks of 8 subjects. The two diets will be consumed for 4 weeks and separated by a 2- to 4-week washout period.

During diet phases, all meals and foods will be provided to ensure optimal diet control using a 7-day cyclic menu. The WFPB diet emphasizes low intakes of red and processed meats and high intakes of whole plant-based foods with water as the drink of choice, as per Canada's Food Guide. The SAD diet reflects current dietary intakes of the French-Canadian adult population in terms of foods, nutrients, and diet quality, as characterized in recent surveys conducted in an age- and a sex-representative sample of adults from the Province of Quebec. An experienced food technician will prepare the diets. Each food and ingredient will be weighed with a precision of ±0.1 g.

During the diet phases, participants will visit the INAF clinical research unit three times weekly (Monday, Wednesday, Friday) to collect their meals and had the option to eat on-site under supervision. At that time, they will also be given their evening meals and the next day's packaged breakfast to take home. Weekend meals will be provided at the Friday visits. A checklist will be provided to all participants to identify the consumed foods. Alcohol, vitamin supplements, and natural health products will not be allowed. Tea and coffee (black) will be allowed (≤2 servings/day without daily fluctuations). Participants will be instructed to maintain their usual physical activity level. At the end of each diet, fasting plasma samples will be collected in ethylenediaminetetraacetic acid (EDTA) tubes. Parts of the samples will be stored at -80℃ for future ancillary analyses. Participants' anthropometry, body composition (DEXA scan), and blood pressure will be measured. To incorporate gender aspects associated with the intervention in knowledge transfer activities, subjects' appreciation of the diets and appetite sensation will be assessed using visual analog scales filled after each meal on day 7 and 28 of each diet.

Objective 1: To investigate the impact of a whole food plant-based diet low in red and processed meats and high in plant foods in place of a standard North American diet on LDL-C concentrations - the primary treatment target in HeFH management. This objective will output a convincing demonstration of the cholesterol-lowering effects of diet in adults with HeFH, supporting the effectiveness of dietary interventions in HeFH management. Investigators will compare post-diet LDL-C levels (primary outcome) using mixed models for repeated measures.

The following analyses will complement those on LDL-C in order to obtain a comprehensive perspective on the impact of diet on CVD risk factors and CVD risk. We will also compare post diet levels in: ApoB; Total cholesterol; Lp(a)-corrected LDL-C; HDL-cholesterol; Triglycerides; Non-HDL-C; ApoA1; Lp(a); C-reactive protein; Fasting plasma glucose; Fasting insulin; HbA1c.

All these parameters will be measured from the plasma samples collected at the end of each diet. We will also compare post-diet systolic and diastolic blood pressure, and compare post-diet ten-year risk of CVD event, using the validated FH risk score. The same statistical approaches as those used for LDL-C will be used for these analyses.

To maximize the study contribution, the following exploratory analyses will be conducted from the per-protocol dataset, to minimize the risk of confounding due to protocol deviations. All of these should be considered exploratory outcomes.

1. Investigators will assess whether diet could influence HeFH detection, given that none of the participants were using cholesterol-lowering medication during the dietary intervention, by comparing the proportion of participants whose post-diets LDL-C levels will exceed the thresholds for FH investigation defined in the Simplified Canadian Definition for FH (≥4.50 mmol/L for 18 to 40 years, and >5.00 mmol/L for over 40 years). Post-diet proportions will be compared with McNemar's test.
2. Investigators will assess the impact of the diets on fasting appetite hormones (total GLP-1 and peptide YY), PCSK9 and noncholesterol sterols, using linear mixed models, as described for LDL-C.
3. To identify the determinants of the LDL-C response to the experimental diets, investigators will evaluate a series of potential determinants using simple linear regression models. The tested determinants will include:

   i. unmodifiable factors (sex, age, LDLR genotype); ii. lifestyle-related factors (BMI, as a surrogate of energy balance51, and mean calorie intake); iii. cardiometabolic health surrogates (CRP, HOMA-IR, total fasting GLP-1, systolic blood pressure); iv. and cholesterol and lipoprotein-metabolism related factors (lathosterol/cholesterol ratio, campesterol/cholesterol ratio, and levels of PCSK9, Lp(a) and LDL-C).

   For all potential determinants, investigators will use values obtained at the end of the control diet to simulate the metabolic state of individuals before adopting a healthy diet. To determine which factors are the most strongly associated with the LDL-C response to the diet, investigators will fit all possible reduced models. The model with highest adjusted R2 - the model with the best balance between goodness-of-fit and complexity - will be selected for presentation. The LDL-C response will be defined as the percent difference between post diet levels and will be treated as the dependent variable. Each potential predictor will be treated as the independent variable. These analyses will be repeated on ApoB response.
4. To support the translation of the findings into clinical practice, investigators will compare the impact of the diets on perceived appetite sensations and meal appreciation, at the end of each diet, using linear mixed models. Diet will be treated as a fixed effect, while subjects will be treated as a random effect. However, we will use an a priori sex-specific approach, motivated by findings from a previous study that reported marked differences between males and females in appetite sensations and diet appreciation following a Mediterranean diet. This sex-specific analysis is intended to maximize the potential for clinical translation, regardless of sex. Thus, the models will include an interaction term. In addition, the models will be adjusted for meal, weekday, daily energy intake, age, BMI, and diet sequence.
5. Investigators will evaluate changes in appetite sensations and meal appreciation between the first and last weeks of each dietary intervention, to understand how repeated exposure to the diets influences these parameters and support the translation of our findings into clinical practice. Again, an a priori sex-specific approach will be used for the aforementioned reasons. For these analyses, assessment period (first week vs last week) will be treated as a fixed effect and participants will be treated as a random effect. To determine the difference between the dietary interventions, an interaction term (assessment period * diet) will be added to the models. Two different models will be fitted according to sex. To assess how sex impacts time-related changes between the two diets, linear mixed models will be used. These models will consider the changes in appetite sensations from the first to the final week of the interventions as the dependent variable. Additionally, an interaction term between sex and diet will be included in the models to examine how the time-related effect of diet on appetite sensations might vary by sex. All these models will be adjusted for meal, weekday, daily energy intake, age, BMI, and sequence.

Objective 2: To assess the impact of a diet low in red and processed meats and high in plant foods in place of a standard North American diet on the plasma metabolome. This objective serves a dual purpose as it will: 1. inform on the dietary impact on systemic metabolism, beyond its impact on LDL-C levels, further supporting the importance of healthy dietary habits in HeFH; and 2. allow the identification of an unbiased HeFH-specific plasma metabolomic signature of a diet low in red and processed meats and high in plant foods to be used as an objective proxy of diet adherence. To document post-diet differences in plasma metabolome (secondary outcome) and identify the metabolomic signature of the WFPB diet, investigators will derive a reproducible multi-metabolite model discriminating the post-WFPB/post-SAD metabolomic profiles.

Objective 3: To evaluate the association between the plasma metabolomic signature of a diet low in red and processed meats and high in plant foods and cardiovascular disease risk. The metabolomic signature will allow to infer how objective adherence to a healthy diet is associated with cardiovascular disease risk in a distinct, large cohort of free-living adults with HeFH. This will provide an innovative demonstration of the role of diet in long-term cardiovascular disease prevention in adults with HeFH, further supporting the importance of a healthy diet in this high-risk population. To evaluate the association between the plasma metabolomic signature of the healthy WFPB diet and cardiovascular disease risk in adults with HeFH, investigators will leverage a distinct cross-sectional cohort of adults with HeFH. Upon recruitment, participants underwent a complete clinical assessment and fasting blood samples were collected in EDTA tubes. Investigators will fit and standardize the WFPB multi-metabolite model (signature) to the cohort metabolomic data. The relationship between the WFPB multi-metabolite model (independent variable) and cardiovascular disease risk factors (plasma lipids, blood pressure, plasma glucose, insulin, HbA1c) will be assessed using linear regressions.

Results will fill key gaps on the short- and long-term influence of diet on cardiovascular health in HeFH.

ELIGIBILITY:
Inclusion criteria:

* Genetically-defined HeFH
* Premenopausal women with a regular menstrual cycle for >3 months
* Postmenopausal women (without hormone replacement)

Exclusion criteria:

* Any cardiovascular disease-risk exacerbating conditions (age >60 years, homozygous FH, personal history of cardiovascular disease, diabetes/anti-diabetic drug use, severe obesity, unstable body weight for >3 months, uncontrolled hypertension, genetic hypertriglyceridemia),
* Allergies/aversions to components of the experimental diets
* Any condition that would interfere with optimal participation in the intervention.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Post-diet differences in LDL-C levels. | This analysis will compare LDL-C levels from plasma samples collected at the end (day 28) of each diet.
  Investigators will compare the impact of a diet low in red and processed meats and high in plant foods in place of a standard North American diet on LDL-C concentrations among adults with HeFH.

SECONDARY OUTCOMES:
Post-diet differences in plasma metabolomics profiles. | This analysis will compare metabolomic profiles from plasma samples collected at the end (day 28) of each diet.
  Investigators will assess the impact of a diet low in red and processed meats and high in plant foods in place of a standard North American diet on the plasma metabolomics profiles to identify the metabolomic signature of the CFG diet. Plasma metabolites will be measured using 3 complementary liquid chromatography-tandem mass spectroscopy methods for 1) polar metabolites (e.g. amino acids), 2) lipids, and 3) free fatty acids.

OTHER OUTCOMES:
Post-diet differences in other atherogenic lipoproteins and lipids | This analysis will compare levels of atherogenic lipoproteins and lipids measured from plasma samples collected at the end (day 28) of each diet
  Investigators will compare the impact of a diet low in red and processed meats and high in plant foods in place of a standard North American diet on plasma levels of atherogenic lipoproteins and lipids (apolipoprotein B, non-HDL-cholesterol, total-cholesterol, triglycerides, lipoprotein(a)).
Post-diet differences in other lipoproteins and lipids | This analysis will compare levels of other lipoproteins and lipids measured from plasma samples collected at the end (day 28) of each diet
  Investigators will compare the impact of a diet low in red and processed meats and high in plant foods in place of a standard North American diet on plasma levels of other lipoproteins and lipids (apolipoprotein A1, HDL-cholesterol).
Post-diet differences in fasting plasma glucose | This analysis will compare levels of fasting plasma glucose (mmol/L) measured from plasma samples collected at the end (day 28) of each diet.
  Investigators will compare the impact of a diet low in red and processed meats and high in plant foods in place of a standard North American diet on fasting plasma levels of glucose (mmol/L).
Post-diet differences in fasting plasma insulin | This analysis will compare levels of insulin (pmol/L) measured from plasma samples collected at the end (day 28) of each diet.
  Investigators will compare the impact of a diet low in red and processed meats and high in plant foods in place of a standard North American diet on fasting plasma levels of insulin (pmol/L).
Post-diet differences in glycated hemoglobin (HbA1c) | This analysis will compare levels of glycated hemoglobin (HbA1c) (%) from plasma samples collected at the end (day 28) of each diet.
  Investigators will compare the impact of a diet low in red and processed meats and high in plant foods in place of a standard North American diet on glycated hemoglobin (HbA1c) (%).
Post-diet differences in systolic and diastolic blood pressure | This analysis will compare systolic and diastolic blood pressure (mm Hg) measured at the end (day 28) of each diet.
  Investigators will compare the impact of a diet low in red and processed meats and high in plant foods in place of a standard North American diet on systolic and diastolic blood pressure (mm Hg).
Post-diet differences in C-reactive protein levels. | This analysis will compare C-reactive protein levels (mg/L) measured at the end (day 28) of each diet.
  Investigators will compare the impact of a diet low in red and processed meats and high in plant foods in place of a standard North American diet on C-reactive protein levels (mg/L).
Post-diet differences in 10-year risk of atherosclerotic cardiovascular disease | This analysis will compare 10-year risk of atherosclerotic cardiovascular disease (%) measured at the end (day 28) of each diet.
  Investigators will compare the impact of a diet low in red and processed meats and high in plant foods in place of a standard North American diet on 10-year risk of atherosclerotic cardiovascular disease (%).
Post-diet difference in HeFH detection. | This analysis will compare the proportion of participants whose post-diets LDL-C levels will exceed the thresholds for FH detection at the end (day 28) of each diet
  Investigators will assess whether diet could influence HeFH detection, given that none of the participants will be using cholesterol-lowering medication during the dietary intervention, by comparing the proportion of participants whose post-diets LDL-C levels will exceed the thresholds for FH investigation defined in the Simplified Canadian Definition for FH (≥4.50 mmol/L for 18 to 40 years, and >5.00 mmol/L for over 40 years). Post-diet proportions will be compared with McNemar's test
Post-diet differences in appetite hormone (total GLP-1, peptide YY) levels. | This analysis will compare total GLP-1 and PYY levels from plasma samples collected at the end (day 28) of each diet.
  Investigators will compare the impact of a diet low in red and processed meats and high in plant foods in place of a standard North American diet on plasma levels of total GLP-1 and peptide YY (PYY) among adults with HeFH.
Post-diet differences in plasma PCSK9 levels | This analysis will compare PCSK9 levels from plasma samples collected at the end (day 28) of each diet.
  Investigators will compare the impact of a diet low in red and processed meats and high in plant foods in place of a standard North American diet on plasma levels of PCSK9 among adults with HeFH.
Post-diet differences in plasma noncholesterol sterols levels | This analysis will compare noncholesterol sterol levels from plasma samples collected at the end (day 28) of each diet.
  Investigators will compare the impact of a diet low in red and processed meats and high in plant foods in place of a standard North American diet on plasma levels of noncholesterol sterols (desmosterol, lathosterol, lanosterol, campesterol, beta-sitosterol, cholestanol) among adults with HeFH.
Determinants of the LDL-C response to the experimental diets | This analysis will assess the influence of the potential determinants measured at the end (day 28) of the SAD diet on the response of LDL-C, calculated as the difference between post-WFPB and post-SAD LDL-C levels.
  Investigators will evaluate a series of potential determinants of the LDL-C response to the experimental diets. The tested determinants will include : (i) unmodifiable factors (sex, age, LDLR genotype); (ii) lifestyle-related factors (BMI, as a surrogate of energy balance51, and mean calorie intake); (iii) cardiometabolic health surrogates (CRP, HOMA-IR, total fasting GLP-1, systolic blood pressure); and (iv) cholesterol and lipoprotein-metabolism related factors (lathosterol/cholesterol ratio, campesterol/cholesterol ratio, and levels of PCSK9, Lp(a) and LDL-C).
Post-diet differences in appetite sensation | Appetite sensation was measured at the end of the first (day 7) and the last week (day 28) of each diet. Changes between day 28 and day 7 will be calculated and compared between diet.
  Investigators will compare between-diet changes in appetite sensation between the first and the last week of each diet in a gender specific approach. Appetite sensation was measured using visual analog scale at the end of the first (day 7) and the last week (day 28) of each diet. Changes between day 28 and day 7 will be calculated and compared between diet.
Association between the plasma metabolomic signature of the healthy CFG diet and LDL-C levels | This analysis will leverage metabolomic profiles from plasma samples collected at the end (day 28) of each diet, but it is not part of the intervention time frame per se.
  Investigators will evaluate the association between the plasma metabolomic signature of the CFG diet (outcome 2) and LDL-C levels (mmol/L) in a cross-sectional cohort of 400 adults with HeFH. The main independent variable will be the CFG multi-metabolite signature which will be modeled as a continuous variable using a z-score. The z-score reflects adherence to the CFG diet (higher z-scores indicate higher adherence to the CFG diet. LDL-C levels (mmol/L) (continuous variables) will be treated as the dependent variable in the linear regression models.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Drouin-Chartier, Study Director — Laval University
Locations (1):
- Institute on nutrition and functional foods, Laval University, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Access to the minimum dataset necessary to interpret, verify, and extend the research reported in this article will be made available upon request through a custom proprietary repository, in accordance with the conditions set by the local ethics review committee on data sharing. Data access requests should be directed to the study investigators.